CLINICAL TRIAL: NCT05961215
Title: IIT2023-03-Vescio-ColdCap: Scalp Cooling to Prevent Hair Loss in Patients Undergoing Stem Cell Transplantation for Multiple Myeloma
Brief Title: Scalp Cooling to Prevent Hair Loss in Patients Undergoing Stem Cell Transplantation for Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Penguin Cold Caps (Unknown)
Responsible Party: Principal Investigator, Robert Vescio, MD, Medical Director, Multiple Myeloma and Amyloidosis Program, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2023-03-Vescio-ColdCap
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Penguin Cold Cap (Experimental): Patients will receive Penguin cold cap: 60 minutes prior to melphalan infusion and continue for 5 hours after melphalan infusion start time, for a total of 6 hours, on Days -2 and -1.
  Interventions: Device: Penguin Cold Cap

INTERVENTIONS:
Device: Penguin Cold Cap — Penguin cold cap: administered 60 minutes prior to melphalan infusion and continue for 5 hours after melphalan infusion start time, for a total of 6 hours, on Days -2 and -1.

SUMMARY:
This pilot study of scalp cooling with Penguin cold caps will examine the effectiveness of scalp cooling to reduce the development of hair loss in 30 participants with multiple myeloma undergoing high-dose chemotherapy with melphalan and autologous peripheral blood stem cell transplant at Cedars-Sinai Medical Center. The investigators will also assess the potential impact of hair loss versus the discomfort and inconvenience of the scalp cooling procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ECOG performance status ≤2
* Confirmed multiple myeloma diagnosis
* Hair covering ≥75% of scalp on physical exam at screening visit
* Planning to undergo SOC high-dose chemotherapy with melphalan (dose to be used = 140 - 200 mg/m2 (with rounding per CSMC guidelines)) followed by an autologous peripheral blood stem cell transplant.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Prior or current use of any scalp cooling treatment
* Hair covering < 75% of the scalp on physical exam at screening visit.
* Medical History and Concurrent Diseases: Reynaud's disease, Cold sensitivity, Cold agglutinin disease, Cryoglobulinemia, Cryofibrinogenemia
* Current spinal or neck injury that may interfere with the subject's participation for the full duration of the study, in the opinion of the treating investigator
* Skin conditions such as psoriasis, eczema, malignancy, or other condition on the scalp that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Current use of oxaliplatin
* Current use of any other investigational agents
* Contraindication to melphalan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vescio, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Penguin Cold Cap
Started | 31
Completed | 30
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Penguin Cold Cap
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.43 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 22
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Development of Hair Loss
Description: Change in development of hair loss will be defined as < 50% hair loss (according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAEs) Version 5, Grade 0 or 1) in 75% of patients treated. In CTCAE (Common Terminology Criteria for Adverse Events) version 5.0, alopecia is graded based on the extent of hair loss, with two main grades: Grade 1 (hair loss less than 50%, not obvious from a distance) and Grade 2 (hair loss of 50% or more, readily apparent). Grade 1 alopecia may be manageable with different hairstyles, while Grade 2 typically requires a wig or other camouflage if desired. Additionally, Grade 2 alopecia is more likely to impact a patient's quality of life. Grade 0 indicates that there is no alopecia (no hair loss) reported
Time Frame: Screening (Day 0), Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Penguin Cold Cap
Number analyzed (Participants) | 30
Participants
  Screening: 0 Alopecia | 30
  Screening: 1 Level | 0
  Screening: 2 Level | 0
  Day 30: 1 Level | 4
  Day 30: 0 Alopecia | 26
  Day 30: 2 Level | 0

2. Secondary Outcome: Patient Determined Decision of Scalp Cooling Benefit
Description: Patient determined decision of scalp cooling benefit will be measured by Scalp Cooling Questionnaire, a homegrown scale ranging from no benefit to substantial benefit, with higher scores representing a better outcome.
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Penguin Cold Cap
Number analyzed (Participants) | 29
Participants
  A big effect - 4 | 2
  Not at all | 8
  Somewhat had an effect - 3 | 6
  A little bit - 2 | 13

ADVERSE EVENTS:
Time Frame: Adverse events will be tracked from Day -2 to Follow-up visits (90 days)
Arm/Group | Penguin Cold Cap
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT05961215/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT05961215/ICF_001.pdf